CLINICAL TRIAL: NCT04807738
Title: Effect of Neuroproprioceptive "Facilitation, Inhibition" Physical Therapy Using Virtual Reality on Upper Limb Mobility and Postural Stability in Multiple Sclerosis
Brief Title: Virtual Reality in Physical Therapy in Multiple Sclerosis
Acronym: VIREMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charles University, Czech Republic (Other)
Responsible Party: Principal Investigator, Kamila Řasová, assoc. prof. PhDr.Kamila Řasová, Ph.D., Charles University, Czech Republic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 1983/21+4772/21 (G-21-02)
Record Dates: First submitted 2021-03-16; First posted 2021-03-19 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Multiple Sclerosis
Keywords: multiple sclerosis; virtual reality; hand dexterity; postural stability; physical therapy; coordination; upper limb fine motor skills; motor programme activating therapy; neuroproprioceptive "facilitation, inhibition"; postural control; functional recovery; Demyelinating Autoimmune Disease; Autoimmune Diseases of the Nervous System
MeSH Terms: conditions — Multiple Sclerosis; Inhibition, Psychological; Autoimmune Diseases of the Nervous System

STUDY DESIGN:
Intervention Model Description: A randomized controlled trial. 110 outpatients will be randomized into two interventional groups, one with face-to-face individual neuroproprioceptive "facilitation and inhibition" physical therapy combining key principles of proprioceptive neuromuscular facilitation (PNF) and motor program activating therapy (MPAT). The second arm will place the same therapy, but virtual reality environment. Participants of both groups - active comparator and virtual reality interventional group will undergo 15 hourly therapies, twice a week in a time range of two months. Before and in a week following the last therapy, all participants will be examined by a blinded independent clinician.
Who Masked: Outcomes Assessor
Masking Description: All participants of the study will undergo a clinical examination including a questionnaire survey, led by a blinded independent examiner, who will not have access to intervention documentation. The examiner will see each patient twice, before the first intervention and in follow-up examination in a week following the last therapy. The examiner will be prohibited to talk about the therapy attended. The patients will be informed about the character of the examination and the importance of the most objectivity possible. All therapists can apply both interventions, therefore masking is more efficient.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neuroproprioceptive "facilitation and inhibition" (Active Comparator): ARM 1 - Neuroproprioceptive "facilitation and inhibition" physical therapy combining key principles of proprioceptive neuromuscular facilitation (PNF) and motor program activating therapy (MPAT), with former positive probative evidence on MS and are recommended for MS intervention.
  Interventions: Other: Neuroproprioceptive "facilitation and inhibition"
- Neuroproprioceptive "facilitation and inhibition" in virtual reality (Experimental): ARM 2. Experimental group, neuroproprioceptive "facilitation and inhibition" physical therapy combining key principles of proprioceptive neuromuscular facilitation (PNF) and motor program activating therapy (MPAT) through virtual reality and software inducing and motivating for movement according to principles of proprioceptive neuromuscular facilitation (PNF) and motor program activating therapy (MPAT). We believe that the VR environment might lead to better results due to greater motivation effect, novelty effect, entertainment effect, as well as activating the reward system. We believe the VR might enhance the activation of mirror neurons, it might also activate proprioception. The present physiotherapist is to ensure proper execution of the tasks. The correlation of the two arms of the study should indicate, whether virtual reality and the software used are as effective, or more effective in sustaining the hand motor function and axial stability, than traditionally led therapy.
  Interventions: Device: Neuroproprioceptive "facilitation and inhibition" in virtual reality

INTERVENTIONS:
Device: Neuroproprioceptive "facilitation and inhibition" in virtual reality — The outpatients will be randomized into groups: Individual neuroproprioceptive "facilitation and inhibition" physical therapy combining key principles of proprioceptive neuromuscular facilitation (PNF) and motor program activating therapy (MPAT) in a real environment and the second arm, the same therapy in virtual reality environment. All participants will undergo 15 sessions, 60 minutes each, twice a week in a period of two months.
  The therapy in the interventional group, uses virtual reality and the new software that was developed specifically for inducing and motivating for movement according to principles of proprioceptive neuromuscular facilitation (PNF) and motor program activating therapy (MPAT). The software allows immediate feedback and moreover, movement is corrected by a present therapist. Evaluation of speed and performance quality might be extracted from the software of virtual reality.
  Arms: Neuroproprioceptive "facilitation and inhibition" in virtual reality
Other: Neuroproprioceptive "facilitation and inhibition" — The first arm of the study will undergo physical therapy with physiotherapeutic approach based on neurophysiological principles using proprioceptive neuromuscular facilitation (PNF) and motor program activating therapy (MPAT) approaches. MPAT makes use of particular motor patterns that evolve in postural control development. The repetition of activated programs, a set of stimuli, applied to change the posture with anatomical centration of the joint under various conditions in leading to better support of postural stabilization while seated, while getting up, stepping forward, and standing, in order to teach the patients to use the acquired motor skills automatically in daily life. PNF is a method used for learning effective movement patterns with high biomechanical effectiveness based on repetitive stimulation of cooperating alfa-motoneurons and proprioceptors in muscle, tendons and joint capsules. Therapy will be individualized and led in the standard face-to-face regiment.
  Arms: Neuroproprioceptive "facilitation and inhibition"

SUMMARY:
The randomized controlled trial is aimed to study the efficacy of virtual reality (VR) and its impact on upper limb function and postural stability in people with mild to severe multiple sclerosis (pwMS). The conceptual idea is to compare two kinds of neuroproprioceptive "facilitation and inhibition" physical therapy, first in a real environment and second in virtual reality, in out-patient therapy that will be held in 15 hourly therapies, 2x a week in a period of two months. The efficacy will be assessed by a blinded independent clinical examiner using clinical examination and questionnaire survey before and in a week following the therapeutic intervention. The main focus is on upper limb gross and fine motor skills, trunk stability and stability, and sit to stand stability.

DETAILED DESCRIPTION:
In 60 - 75% of people with multiple sclerosis (MS) an upper limb mobility dysfunction (unilateral or bilateral manual dexterity, sensibility impairment, tremor) is present, resulting in reduced participation in activities of daily living.

Physiotherapy has a crucial impact on upper limb mobility, although there are many approaches applied (exercise/strengthening exercise, endurance training, sensory training, constraint-induced movement therapy, robotic rehabilitation therapy, etc.).

Virtual reality is an innovative technological concept using game mechanisms that facilitate concentration and motivation in task performance. Current research implies that VR is a safe and effective method in gait and balance//stability rehabilitation therapy and with less evidence, for upper limb mobility improvement. It is expected that a greater therapeutic effect is a result of multifactorial sense stimulation and dopamine centres in the brain.

A pilot project showed that virtual reality without the prompt feedback of a physiotherapist is not more effective than standard therapy. A new therapeutic software using virtual reality spontaneously motivating the patient for movement realization was developed in cooperation with the Department of informatics and computer science Faculty of applied sciences University West Bohemia. Accurate execution of neuroproprioceptive "facilitation and inhibition techniques" physical therapy combining key principles from proprioceptive neuromuscular stabilization (PNS) and motor program activating therapy (MPAT), ensures a present physiotherapist. These principles have shown the effect in therapy in pwMS. Participants will be randomized into two arms of the study, both implementing neuroproprioceptive "facilitation and inhibition" physical therapy, first in a real environment and second in VR.

The investigators expect that VR intervention shall improve upper limb motor functions, trunk muscles coordination, improve the performance of activities of daily living and quality of life in pwMS more than identical therapy not using VR.

The effect of both interventions will be assessed using validated tests for clinical examination- Five times Sit to Stand test (5STS), Nine Hole Peg Test (9HPT), Hand Grip Strength (HGS), Box and Block Test (BNB), accelerometer for tremor examination. Validated questionnaires will be used, specifically the Multiple Sclerosis Impact Scale (MSIS-29), EQ-5D-3L health questionnaire, Visual Analogue Scale, and a questionnaire dealing with individual virtual reality intervention evaluation.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria comprise of a definite diagnosis of multiple sclerosis, EDSS score ≥ 2 a ≤ 7 ((10); determined by neurologist), no history of relapse, no history of change in disease-modifying treatment, no history of corticosteroid therapy in the past three months prior to recruitment.

Exclusion Criteria:

* The exclusion criteria include other factors influencing mobility (history of stroke, pregnancy, traumatic injury of limb/s. Severe cardiovascular or orthopedic dysfunction, impaired cognitive functions in the course of examination and/or consecutive therapy.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2025-01-02 (Actual); Study Completion 2025-02-01 (Actual)

PRIMARY OUTCOMES:
Nine Hole Peg Test (9HPT) - change pre/post intervention | Pre-assessment (baseline testing), Post-assessment (immediately in a week following the last procedure)
  The NHPT requires participants to repeatedly place and then remove nine pegs into nine holes, one at a time, as quickly as possible. Lower number (quicker time) means better result.
Box and Block Test (BNB) - change pre/post intervention | Pre-assessment (baseline testing), Post-assessment (immediately in a week following the last procedure)
  The Box and Block Test tests gross manual dexterity. This test consists of moving, one by one, the maximum number of blocks from one compartment of a box to another of equal size, originally, within 60 seconds. A lower number (quicker time) means better result.
Hand Grip Strength (HGS) -change pre/post intervention | Pre-assessment (baseline testing), Post-assessment (immediately in a week following the last procedure)
  Jamar Hydraulic Hand Dynamometer measures isometric grip force and strength. The higher value, the better function (higher strength).
Tremor; Frequency for which the smoothed power spectral density is maximal (fMAX) | Pre-assessment (baseline testing), Post-assessment (immediately in a week following the last procedure)
  The spectral characteristic of postural tremor measured by the 3-axis accelerometer and 3-axis gyroscope chip (Motion Tracking sensor MPU-6050) - lower value, lower tremor.
Tremor; Power of the signal in band from f1 to f2 (Pf1-f2) | Pre-assessment (baseline testing), Post-assessment (immediately in a week following the last procedure)
  The spectral characteristic of postural tremor measured by the 3-axis accelerometer and 3-axis gyroscope chip (Motion Tracking sensor MPU-6050) - lower value, lower tremor.
Five times Sit to Stand test (5STS) -change pre/post intervention | Pre-assessment (baseline testing), Post-assessment (immediately in a week following the last procedure)
  The test assesses time when people stand and sit repeatedly five times. The lower the time to complete the test the better the outcome of the test.

SECONDARY OUTCOMES:
Multiple Sclerosis Impact Scale (MSIS-29) - change pre/post intervention | Pre-assessment (baseline testing), Post-assessment (immediately in a week following the last procedure)
  A 29-item self-report measure with 20 items associated with a physical scale and 9 items with a psychological scale. Items ask about the impact of MS on a day-to-day life in the past two weeks. All items have 5 response options: 1 "not at all" to 5" extremely". Each of the two scales is scored by summing the responses across items, then converting to a 0-100 scale where 100 indicates the greater impact of the disease on daily function (worse health).
EQ-5D-3L-health questionnaire - change pre/post intervention | Pre-assessment (baseline testing), Post-assessment (immediately in a week following the last procedure)
  Descriptive system for health-related quality of life states in adults, consisting of five dimensions (Mobility, Self-care, Usual activities, Pain & discomfort, Anxiety & depression), each of which has three severity levels that are described by statements appropriate to that dimension. A higher number means a worse quality of life.

OTHER OUTCOMES:
Kinematic analysis | Pre-assessment (baseline testing), Post-assessment (immediately in a week following the last procedure)]
  The kinematic data from the HCT vive VR and the VR software will be available for the intervention and the control group to evaluate performance i regarding accuracy (spatial distance in meters).
Functional Magnetic Resonance Imaging | Pre-assessment (baseline testing), Post-assessment (immediately in a week following the last procedure)]
  MR examination (E1 and E2) will include measurements of functional stimulated data related to motoric inputs, functional connectivity measurement (resting state measurement, individually assessed), structural images (three-dimensional SPACE (sampling perfection with application-optimized contrasts using different flip angle evolutions) FLAIR (fluid-attenuated inversion recovery) and three-dimensional magnetisation prepared-RApid gradient echo (3D MP-RAGE)) and structural connectivity, with 106 spatial directions and 3b-factors allowing the reconstruction not only of fractional anisotropy but also the diffusion kurtosis maps
MR tractography and Diffusion-Weighted Imaging | Pre-assessment (baseline testing), Post-assessment (immediately in a week following the last procedure)]
  MR scans will be performed according to an optimized protocol for diffusion-weighted imaging (DWI) using a spin-echo echo-planar imaging (SE-EPI) sequence; repetition time (TR) = 4500 ms, echo time (TE) = 92 ms, 69 axial slices, field of view (FOV) = 200 mm, 106 diffusion directions, and a voxel size of 2 × 2 × 2 mm³. A multishell diffusion scheme with b-values of 0, 1000, and 3000 s/mm² will be employed for baseline and follow-up scans. DWI provides insights into the microstructural integrity of brain tissue by highlighting areas where diffusion is restricted.
  To compare longitudinal changes in white matter tracts differential tractography will be performed. MR tractography visualizes neural pathways by mapping the direction of water diffusion along white matter tracts, helping to understand brain anatomy and connectivity. The aim of these techniques is to study brain structure and function in relation to the PT intervention.
Monocyte-Derived Dendritic Cells | Pre-assessment (baseline testing), Post-assessment (immediately in a week following the last procedure)]
  From a sample of peripheral blood (K3EDTA tubes), peripheral blood mononuclear cells will be isolated. Monocytic cell fraction will be cultivated of adherent monocytes supplemented with human granulocyte-macrophage colony-stimulating factor and human interleukin. CD cell markers will be analyzed on leukocytes and MoDC: CD3, CD19, CD4, CD8, CD25, CD127, CD279, CD122, CD14, CD16, CD33, CD64, CD86, CD11c, HLA-DR, CD63 on flow cytometer using anti-human monoclonal antibodies, results in %.
Analysis of Long Non-Coding RNA (real-time Quantitative PCR) | Pre-assessment (baseline testing), Post-assessment (immediately in a week following the last procedure)]
  From a peripheral blood sample in 10ml K3EDTA test tube RNA will be isolated using the NucleoSpin RNA Midi blood Mini, according to the manual. Total RNA (1μg) is converted into cDNA using standard protocol procedures and reagents (Thermo Fischer Scientific, Waltham, MA, USA).The study will include an analysis of preselected long non-coding RNA (MALAT1, MEG3, H19, GAS5, PARTICLE, TINA) determined by quantitative PCR. For normalization purposes and relative gene expression analysis, endogenous control genes are assessed (GAPDH, B2M). Measured in a StepOne Real-time PCR system instrument (VWR, Prague). All samples will be measured in triplets. Relative gene expression is quantified using the 2(-ΔΔCt) method.

CONTACTS AND LOCATIONS:
Overall Officials: Kamila Rasova, as.prof.Dr., Study Director — Clinic of rheumatology and rehabilitation,Third medical faculty CU and Faculty Thomayer Hospital
Locations (2):
- Czechia (2):
  - Department of neurology, Prague
  - Deparment of revmatology and rehabilitation, Prague

IPD SHARING:
Plan to Share IPD: No
Only anonymised data will be made available to other researchers on reasonable request.

REFERENCES:
- [Derived] Miznerova B, Reissigova J, Vasa L, Frank J, Hudec M, Rodina L, Herynkova A, Havlik J, Tintera J, Rydlo J, Ibrahim I, O'Leary VB, Cerna M, Jurickova I, Pokorna M, Philipp T, Hlinovska J, Stetkarova I, Rasova K. Virtual reality-based neuroproprioceptive physiotherapy in multiple sclerosis: a protocol for a double-arm randomised assessor-blinded controlled trial on upper extremity function, postural function and quality of life, with molecular and functional MRI assessment. BMJ Open. 2025 Jan 9;15(1):e088046. doi: 10.1136/bmjopen-2024-088046. PMID 39788766